CLINICAL TRIAL: NCT01404104
Title: A Pilot Study of Neo-adjuvant Temsirolimus in Patients With Advanced Renal Cell Carcinoma Undergoing Definitive Therapy With Radical Nephrectomy, or Cytoreductive Nephrectomy: Analysis if Serum and Tissue Biomarkers
Brief Title: Neo-adjuvant Temsirolimus in Patients With Advanced Renal Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Collaborators: McMaster University (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Anil Kapoor, MD, FRCSC, St. Joseph's Healthcare Hamilton
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIS-003-09
Record Dates: First submitted 2011-07-19; First posted 2011-07-27 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Temsirolimus (pre-surgery) (Experimental)
  Interventions: Drug: Temsirolimus (pre surgery)

INTERVENTIONS:
Drug: Temsirolimus (pre surgery) — Temsirolimus will be given to patients 12 weeks prior to surgery (with a one week off period right before the surgery date).
  Other Names: Temsirolimus

SUMMARY:
Temsirolimus is a drug that is being studied to possibly treat kidney cancer. It works by starving the cancer of nutrients, by cutting off the blood supply, which is hoping to shrink the cancer. This study will look at the experimental use of temsirolimus, 12 weeks prior to the surgical removal of the entire kidney or a portion of the kidney that is involved by the tumor.

DETAILED DESCRIPTION:
This study will also find out whether or not there are certain biological factors that show up in patients during their treatment with this drug. This will be able to predict how their disease will respond to the therapy (biomarkers), and this will possibly allow anti-cancer therapies to be developed in the future to tailor to a patient's needs.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old and capable of giving informed consent.
* Patient has radiological evidence of RCC consisting of: CT scan with stage T2, T3, T3a, T4, or any stage T with N1/2 and/or metastatic disease.
* Patient is already having a nephrectomy.
* Adequate cardiac function as assessed by electrocardiogram (ECG).
* Patient is will to have a kidney biopsy at baseline/screening.
* Patient has scored a 0 or 1 on the ECOG.
* Patient is negative for HIV, Hepatitis B, Hepatitis C
* If patient is a woman of child-bearing potential, they have to have a negative pregnancy test.

Exclusion Criteria:

* Patient has stage T1 disease without metastases.
* Patient has abnormal laboratory values at screening within the following ranges:
* Absolute neutrophil count ≤1.5 x 10(9)/L; Platelet count ≤ 100 x 10(9)/L
* Leukocyte count ≤ 3 x 10(9)/L; Hemoglobin ≤ 80 g/L
* Serum creatinine ≥ 2.0 x the upper normal limit (UNL)
* Total bilirubin ≤ 1.5 x UNL; AST and ALT ≤ 3.0 x UNL
* Fasting serum cholesterol ≤ 9.0 mmol/L
* Fasting serum triglycerides ≤ 5.0 mmol/L
* Patients with a known hyper-sensitivity to Temsirolimus.
* Other currently active malignancies.
* Currently taking any medications known to interfere with the metabolism of Temsirolimus.
* Patients receiving anticoagulation with warfarin.
* Patients with a history of pulmonary hypertension or interstitial lung disease.
* Unstable angina as judged by the primary investigator, or any recent MI in the last 180 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
The rate of change in response of primary tumor and metastases (if applicable)in participants. | Baseline, Weeks 1-12, follow up every 3 months for years 1 and 2, and every 6 months for following three years (5 years in total).
  Rate of Change in response of primary tumor and metastases (if applicable) to neo-adjuvant Temsirolimus in terms of tumour size and appearance (RECIST imaging response criteria) as determined by CT or MRI.

SECONDARY OUTCOMES:
Average time for disease progression. | At every visit; baseline, weekly visits, and follow-up.
  Patients will be seen at baseline and 12 weeks prior to surgical removal of the entire kidney or a portion of the kidney involved by tumour. If there has been metastases then patients might remain on the study treatment with temsirolimus following the surgery, for a maximum of 24 months or until disease progression. The total duration of the study is up to 5 years.
Quality of life data | Baseline, weekly visits, follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Anil Kapoor, MD, Principal Investigator — McMaster Institute of Urology - St. Joseph's Healthcare Hamilton
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada